CLINICAL TRIAL: NCT04979780
Title: Observational Studies in Cancer Associated Thrombosis for Rivaroxaban - United States Cohort
Acronym: OSCAR-US
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21982
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Treatment of Venous Thromboembolism in Cancer Patients; Prophylaxis of Recurrent Venous Thromboembolism in Cancer Patients
MeSH Terms: interventions — Rivaroxaban; Heparin, Low-Molecular-Weight; N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients with acute venous thromboembolism (VTE): Cancer-associated thrombosis (CAT) patients treated with Rivaroxaban or any DOAC (Direct Oral Anticoagulants) or LMWH (Low molecular weight heparin).
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Low molecular weight heparin (LMWH); Drug: Direct Oral Anticoagulants (DOAC)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Retrospective cohort analysis using US Optum De-Identified EHR data.
Drug: Low molecular weight heparin (LMWH) — Retrospective cohort analysis using US Optum De-Identified EHR data. LMWH (dalteparin, enoxaparin, tinzaparin)
Drug: Direct Oral Anticoagulants (DOAC) — Retrospective cohort analysis using US Optum De-Identified EHR data. DOAC (apixaban, dabigatran, edoxaban, rivaroxaban).

SUMMARY:
Patients with active cancer are ~5-fold more likely to develop a venous thromboembolism (VTE) than those without. When VTE occurs, cancer patients carry an up to a 3-fold higher rate of thrombosis recurrence and ~twice the risk of bleeding during anticoagulation. Therefore, it is critical to utilize anticoagulants that optimize efficacy while minimizing bleeding risk when treating cancer-associated thrombosis (CAT).

Guidelines list direct-acting oral anticoagulants (DOACs) as an alternative to low molecular-weight heparin (LMWH) for treatment of CAT. The strength-of-recommendation for DOACs is based on data from multiple randomized controlled trials (RCTs) comparing them to LMWHs to treat CAT, with results suggesting DOACs may reduce thrombosis risk but with potentially more frequent bleeding (particularly in those with certain gastrointestinal and genitourinary cancers).

Observational studies evaluating DOACs for CAT treatment have been published, but these studies have been either single-arm, evaluated cancer subtypes not recommended for DOAC treatment, were of limited sample size and/or employed heterogeneous definitions of active cancer. We seek to evaluate the effectiveness and safety of rivaroxaban versus LMWH for CAT treatment in active cancer patients using a large de-identified electronic health record database.

Retrospective cohort analysis using US Optum® De-Identified EHR data. We will use Optum EHR (electronic health records) data from November January 1, 2012 through latest available data (currently September 2020).

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years of age at the time of anticoagulation initiation.
* Have active cancer admitted to the hospital, emergency department or observation unit for acute DVT and/or PE.
* Treated with rivaroxaban (or any DOAC in secondary analysis) or LMWH as their first anticoagulant on day 7 post-acute CAT event diagnosis (index date) o increase the probability of accurately classifying patients' intended outpatient anticoagulant for CAT treatment and that patients are compared at the same point from diagnosis.
* Have been active in the data set for at least 12-months prior to the index event (based on the "First Month Active" field) and had at least one provider visit in the 12-months prior to the acute VTE event (baseline period).

Exclusion Criteria:

* Evidence of atrial fibrillation, recent hip/knee replacement (within 35 days of index VTE), ongoing VTE treatment, valvular heart disease defined as any rheumatic heart disease, mitral stenosis, or mitral valve repair/replacement.
* Pregnancy.
* Initiation of rivaroxaban at a dose other than 15 mg twice daily or non-therapeutic doses of other DOAC or LMWH (e.g., enoxaparin at a dose other than 1 mg/kg twice daily or 1.5 mg/kg once daily; dalteparin at a dose other than 200 IU/kg of total body weight)
* Evidence of use of anticoagulation use during the 12-months prior per written prescription or patient self-report

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The Optum EHR database includes longitudinal patient-level medical record data for ~91+ million patients seen at ~700+ hospitals and ~7,000+ clinics across the US. The study population of interest will be patients with cancer, admitted to the hospital, emergency department or observation unit for acute DVT and/or PE on or after January 1, 2013 (to correspond with the US availability of rivaroxaban for VTE treatment), being treated with rivaroxaban (or any DOAC in secondary analysis) or LMWH on day 7 post-acute VTE diagnosis (index date), and have been active in the data set for at least 12-months prior to the index event (based on the "First Month Active" field) and had at least one provider visit in the 12-months prior to the acute VTE event (baseline period).
Sampling Method: Non-Probability Sample
Enrollment: 3708 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Risk of recurrent VTE | at 3 month after treatment
Any clinically-relevant bleeding-related hospitalization | at 3 month after treatment
  Cunningham algorithm for identification of bleeding-associated hospitalizations
All-cause mortality | at 3 month after treatment

SECONDARY OUTCOMES:
Recurrent VTE at 6- and 12-months post-index VTE | at 6 and 12 months post-index VTE
Composite of any major or clinically-relevant nonmajor bleeding-related hospitalization at 6- and 12-months post-index VTE | at 6 and 12 months post-index VTE
  including:
  * Intracranial hemorrhage (ICH)
  * Critical organ bleeding (e.g., intracranial, intraspinal, intraocular, retroperitoneal, intraarticular, or pericardial bleeding or intramuscular with compartment syndrome)
  * Extracranial bleeding-related hospitalizations
Any clinically-relevant bleeding-related hospitalization | at 6 and 12 months
  per the Cunningham algorithm for identification of bleeding-associated hospitalizations
Intracranial hemorrhage (ICH) | at 3, 6 and 12 months
Critical organ bleeding | at 3, 6 and 12 months
Extracranial bleeding-related hospitalizations | at 3, 6 and 12 months
All-cause mortality at 6- and 12-months. | at 6 and 12 months
Incidence rates of recurrent VTE | at 3, 6 and 12 months
  Incidence rates of recurrent VTE in DOAC and LMWH patients experiencing CAT regardless of the bleeding risk associated with cancer type.
Incidence rates any clinically-relevant bleeding-related to recurrent VTE | at 3, 6 and 12 months
  Incidence rates of any clinically-relevant bleeding-related in DOAC and LMWH patients experiencing CAT regardless of the bleeding risk associated with cancer type.
All cause-mortality | at 3, 6 and 12 months
  Incidence rates of all cause-mortality in DOAC and LMWH patients experiencing CAT regardless of the bleeding risk associated with cancer type.
Duration of anticoagulation treatment | at 3, 6 and 12 months
DOAC discontinuation rates at 3-, 6- and 12-months follow-up | at 3, 6 and 12 months
LMWH discontinuation rates at 3-, 6- and 12-months follow-up | at 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Background] Caroti KS, Becattini C, Carrier M, Cohen AT, Ekbom A, Khorana AA, Lee AYY, Brescia C, Abdelgawwad K, Psaroudakis G, Rivera M, Schaefer B, Brobert G, Coleman CI. Rivaroxaban versus Apixaban for Treatment of Cancer-Associated Venous Thromboembolism in Patients at Lower Risk of Bleeding. TH Open. 2023 Jul 10;7(3):e206-e216. doi: 10.1055/s-0043-1770783. eCollection 2023 Jul. PMID 37435565
- [Derived] Coleman CI, Caroti KS, Abdelgawwad K, Psaroudakis G, Fatoba S, Rivera M, Schaefer B, Brobert G, Khorana AA, Becattini C, Lee AYY, Ekbom A, Carrier M, Brescia C, Cohen AT. Effectiveness and Safety of Rivaroxaban and Low Molecular Weight Heparin in Cancer-Associated Venous Thromboembolism. JACC CardioOncol. 2023 Feb 7;5(2):189-200. doi: 10.1016/j.jaccao.2022.10.014. eCollection 2023 Apr. PMID 37144109
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/21982